CLINICAL TRIAL: NCT06831825
Title: A Phase I Study of Safety and Preliminary Efficacy of YAP101 in Subjects With Ischemic Heart Failure and Reduced Ejection Fraction
Brief Title: Study Assessing Left Ventricular Administration of a Genetic Medicine Directing Organ Regeneration in Heart Failure
Acronym: SALVADOR-HF
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: YAP Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YAP101-C001
Record Dates: First submitted 2025-01-23; First posted 2025-02-18 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: YAP101; YAP Therapeutics; YAPtx; AAV; Regenerative medicine; Cardiac regeneration; heart regeneration; gene therapy; shRNA; gene silencing; tissue renewal; cardiac repair; heart failure; HFrEF; HF; Heart failure with reduced ejection fraction; NYHA
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Cohort 1: 5e12 vg YAP101 (Experimental): 3 to 6 subjects
  Interventions: Combination Product: YAP101 (AAV9-Sav-shRNA)
- Cohort 2: 1e13 vg YAP101 (Experimental): 3 to 6 subjects
  Interventions: Combination Product: YAP101 (AAV9-Sav-shRNA)
- Cohort 3: 5e13 vg YAP101 (Experimental): 3 to 6 subjects
  Interventions: Combination Product: YAP101 (AAV9-Sav-shRNA)
- Cohort 4 (Dose Level Expansion): Dose level TBD (Experimental): Up to 6 subjects
  Interventions: Combination Product: YAP101 (AAV9-Sav-shRNA)

INTERVENTIONS:
Combination Product: YAP101 (AAV9-Sav-shRNA) — YAP101 delivered using YAPCATH-101

SUMMARY:
This clinical trial investigates the safety and preliminary effectiveness of YAP101, a gene therapy designed to improve heart function in adults with ischemic heart failure and reduced ejection fraction (HFrEF). Ischemic heart failure, often resulting from a prior heart attack, leads to poor heart function and quality of life. Current treatments are limited, and there is an urgent need for new therapies.

YAP101 works by delivering a gene therapy using a specialized vector to heart cells, targeting a pathway involved in heart repair. By temporarily activating heart muscle regeneration, YAP101 aims to restore damaged tissue, reduce scarring, and improve the heart's pumping ability.

The study will enroll participants who will receive a one-time dose of YAP101 via a minimally invasive cardiac injection. Researchers will monitor participants over 12 months to assess safety and changes in heart function, exercise tolerance, and quality of life.

DETAILED DESCRIPTION:
This Phase I, single-center, open-label, dose-escalation trial evaluates the safety, tolerability, and preliminary efficacy of YAP101 in adults with ischemic heart failure and reduced ejection fraction (HFrEF). YAP101, a novel gene therapy, delivers adeno-associated virus with a cardiomyocyte-specific promoter to express short hairpin RNAs (shRNAs) targeting Salvador 1 (SAV1), a key regulator of the Hippo signaling pathway. By transiently suppressing this pathway, YAP101 aims to induce cardiomyocyte regeneration, reduce fibrosis, and improve myocardial function.

Eligible subjects will undergo a one-time transendocardial injection of YAP101 at one of three dose levels (5.0e12, 1.0e13, or 5.0e13 viral genomes/subject) using an investigational cardiac injection catheter. Following administration, subjects will be monitored for safety and functional outcomes through a series of outpatient visits over 12 months. Primary endpoints include the incidence of dose-limiting toxicities, adverse events, and the determination of the maximum tolerated dose (MTD). Secondary endpoints include changes in cardiac function assessed via MRI, biomarkers, exercise tolerance, and quality of life metrics.

Safety will be overseen by an independent Safety Review Team (SRT), which will assess data before dose escalation. The study employs a 3+3 dose-escalation design to identify the MTD while minimizing risks. Subjects who complete the study will have the option to enroll in a long-term follow-up study for up to 5 years.

The trial addresses the significant unmet need for regenerative therapies in heart failure, leveraging preclinical evidence of efficacy and safety. YAP101 has shown promising results in animal models, improving cardiac function, reducing fibrosis, and enhancing myocardial repair without significant adverse effects.

ELIGIBILITY:
Inclusion Criteria:

To participate, a subject MUST:

1. Be ≥ 18 and < 80 years of age;
2. Have medically stable heart failure of ischemic etiology, secondary to MI with NYHA class II or III symptoms for at least 12 months before the initiation of screening procedures;
3. Have a left ventricular ejection fraction (LVEF) ≥ 20% and ≤ 40% by cMRI at screening and baseline;
4. The subject is not a candidate for either percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG) surgery as determined by the principal investigator (or designee) in consultation with an interventional cardiologist during the screening period;
5. Be on stable, outpatient, maximally tolerated guideline directed medical therapy (GDMT) for HF for 6 weeks, unless contraindicated, and remain stable during the screening period;
6. Left ventricular (LV) end diastolic wall thickness of at least 8mm at the potential myocardial site for injection;
7. Be a candidate for cardiac catheterization;
8. Agree to protocol defined requirements for contraception;
9. Provide written informed consent.

Exclusion Criteria:

To participate, a subject MUST NOT HAVE:

1. Valvular heart disease including 1) mechanical or bioprosthetic heart valve; or 2) severe valvular (any valve) insufficiency/regurgitation within 12 months of consent;
2. Aortic stenosis with valve area ≤ 1.5cm2;
3. Prior heart transplant, history of LV reduction surgery, cardiomyoplasty, passive restraint device
4. Had an acute myocardial infarction within the prior 30 days before initiation of screening;
5. Unstable angina pectoris within 30 days before initiation of screening procedures;
6. Idiopathic, valvular, peri/post-partum cardiomyopathy or other cardiomyopathy of non-ischemic etiology;
7. Restrictive, obstructive, or infiltrative cardiomyopathy; pericardial constriction; amyloidosis; or uncorrected thyroid disease;
8. A history of ischemic or hemorrhagic stroke within 90 days of screening;
9. Liver dysfunction, as evidenced by enzymes (e.g., AST, ALT, alkaline phosphatase) greater than 3 times upper limit of normal;
10. A baseline eGFR <35 mL/min/1.73m2;
11. Diabetes with poorly controlled blood glucose levels (HbA1c > 10%);
12. A hematologic abnormality during baseline testing;
13. Coagulopathy (INR > 1.5) not due to a reversible cause (e.g., warfarin and/or Factor Xa inhibitors); Subjects who cannot be withdrawn from anticoagulation will be excluded;
14. An underlying autoimmune disorder or current immunosuppressive therapy;
15. A contrast allergy that cannot adequately be managed by premedication;
16. Received cell-based therapy from any source;
17. Received any viral vector mediated gene therapy;
18. Evidence of active systemic infection at time of study product delivery;
19. HIV and/or active HBV, HCV or Covid-19 infection at screening or baseline;
20. Presence of LV thrombus;
21. Presence of a pacemaker or ICD generator with any of the following limitations/conditions:

    1. manufactured before the year 2000
    2. leads implanted < 6 weeks prior to screening
    3. non-transvenous epicardial leads
    4. subcutaneous ICDs
    5. any other condition that, in the judgment of device-trained staff, would deem an MRI contraindicated;
22. A cardiac resynchronization therapy (CRT) device implanted < 3 months prior to consent;
23. Other MRI contraindications
24. Mobitz II or higher degree atrioventricular block without a functioning pacemaker within 3 months of consent;
25. A history of drug abuse or alcohol abuse, or documented medical, occupational, or legal problems arising from the use of alcohol or drugs within the past 24 months;
26. Cognitive or language barriers that prohibit obtaining informed consent or any study elements;
27. Participation (currently or within the previous 30 days) in a cardiac related investigational therapeutic (including stem cell and gene-based therapies) or device trial;
28. Pregnancy, lactation, plans to become pregnant in the next 12 months, or is unwilling to use acceptable forms of birth control during study participation;
29. Expected survival < 1 year in the judgment of the investigator;
30. Active malignancy within the past 3 years (exceptions: localized prostate cancer, cervical or breast cancer in situ, or nonmelanoma skin cancer that has been definitively treated);

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of the following: DLTs and AEs | 12 months
  Incidence of dose limiting toxicities and adverse events
Maximum tolerated dose | 12 months
  Maximum tolerated dose

SECONDARY OUTCOMES:
Exercise tolerance by six minute walk test (6MWT) | 12 months
  6MWT distance change from baseline in meters
New York Heart Association (NYHA) Classification | 12 months
  NYHA Classification change from baseline (lower values indicate less severe disease, scale from class I to class IV)
Major Adverse Cardiac Events (MACE), including death, MI, revascularization with or without stroke, MACCE | 12 months
  Incidence
Hospitalization for HF and/ or other exacerbation of HF (non-hospitalization) | 12 months
  Incidence
Cumulative days alive and out of the hospital | 12 months
  Days and total days out-of-hospital as a % of total days alive post study intervention
LVEF by cardiac MRI | 12 months
  Change from baseline, %
LVEFI by cardiac MRI | 12 months
  Change from baseline, % per kg
LVEDV by cardiac MRI | 12 months
  Change from baseline, mL
LVEDVI by cardiac MRI | 12 months
  Change from baseline, mL per kg
LVESV by cardiac MRI | 12 months
  Change from baseline, mL
LVESVI by cardiac MRI | 12 months
  Change from baseline, mL per kg
Premature ventricular contraction (PVC) burden | 12 months
  Change from baseline, %
Atrial fibrillation (AFib) burden | 12 months
  Change from baseline, %
BNP (cardiac biomarker) | 12 months
  Change from baseline, %
NT-proBNP (cardiac biomarker) | 12 months
  Change from baseline, %
Health related quality of life as assessed by Minnesota Living with Heart Failure Questionnaire (MLHF) | 12 months
  Change in Score from baseline (lower values indicate higher quality of life, scale from 0-105)
Survival | 12 months
  Days
Cardiac transplant | 12 months
  Incidence
Left ventricular assist device (LVAD) implantation | 12 months
  Incidence
Anti-AAV9 capsid antibodies | 12 months
  Change in titer from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Postalian, MD, Principal Investigator — Texas Heart Institute
Locations (1):
- Texas Heart Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No